CLINICAL TRIAL: NCT04653662
Title: Multi-center, Open-label, Non-randomized, Single-arm Clinical Study to Assess the Safety and Performance of Earol® in Adult Patients With Ear Wax
Brief Title: Earol Madrid Study
Acronym: EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HL Healthcare Ltd (Industry)
Collaborators: AKRN Scientific Consulting, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD1620-001
Record Dates: First submitted 2020-11-16; First posted 2020-12-04 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cerumen Impaction of Both Ears
Keywords: Ear Wax Removal; Ear Wax; Earol; Olive oil; Cerumen; Impaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Treatment group arm. Open label. Only 1 arm study
  Interventions: Device: Earol

INTERVENTIONS:
Device: Earol — Treated with Earol on both ears and subsequent removal after 6 days of application
  Other Names: Ear Wax removal

SUMMARY:
Accumulation of ear wax in the external ear canal is a common pathology. The presence of ear wax not only interferes with the clinician's view of the tympanic membrane, but may also result in hearing loss and vertigo, and may predispose to ear infections.

Removal of ear wax is facilitated using a variety of cerumenolytics, or ear wax solvents. The current study is designed to evaluate the safety and the cerumenolytic effects of the Earol product, when dosed into the auditory canal prior to the dewaxing and ear cleaning procedure. This study is designed to be conducted in the primary care setting as a prospective clinical trial.

A detailed literature review has been conducted to provide a background summary of relevant information on the disease/pathology, other available treatment options and the pre-clinical testing and clinical research that has been conducted to date on the intended population or related populations and/or the device.

The aim for conducting this clinical investigation is to perform a PMCF to evaluate the safety and performance of Earol. Although there are alternative methods for ear wax removal, Earol represents a simple method based on natural ingredients (olive oil) which aids the removal of ear wax as well as prevents appearance of clinical symptoms in the ear canal (E.g. reducing itching and irritation).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to provide written informed consent prior to any clinical investigation related procedure;
* Male or female patients over 18-year-old;
* Presence of ear wax in both ear canals with a minimum of > 50% ear wax blockage in at least one ear (level 4) and > 25% blockage in the contralateral ear (level 3) as assessed using the TMVSS;
* Subject must be willing and able to perform all the visits, follow the PI instructions and complete the follow-up of the study.

Exclusion Criteria:

* Subject is currently participating in another clinical investigation or has participated in another clinical investigation in the past 30 days prior to the start of the present study;
* Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period;
* Presence of other anatomic or comorbid conditions (e.g. ear eczema or seborrhea), or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness;
* Presence or history of a tympanic membrane perforation or tympanostomy tubes at any time during the previous 6 months;
* Presence or history of a known or suspected ear infection (i.e. otitis externa or otitis interna) in the previous 2 months;
* Presence of a known or suspected chronic suppurative otitis media;
* Presence or history of a known or suspected keratosis obturans;
* Presence of known or suspected mastoiditis;
* Use of any ototopical drug or OTC product or ear wax-removal product (except for water or physiologic saline) during the preceding 3 days;
* Hypersensitivity to any product ingredient(s) or history of anaphylactic/anaphylactoid reactions;
* Temporal bone neoplasm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
SAEs and AEs reported | Day 6
  Adverse Events (AEs) and Serious Adverse Events (SAEs) post-treatment

SECONDARY OUTCOMES:
Cerumen blockage assesment | Day 0 and Day 6
  Visualization of the tympanic membrane where cerumen blockage will be assessed post-treatment through the literature and protocol described tool TMVSS (Tympanic Membrane
  Visualization Scoring System). This scale measures the level of obstruction of the ear canal by assessing the level of obstruction when trying to visualize the tympanic membrane with an otoscope.
  Level of obstruction 1 - < 3 % Level of obstruction 2 - 3 - 25 % Level of obstruction 3 - 26 - 50 % Level of obstruction 4 - 51 - 75 % Level of obstruction 5 - 76 - 100 %
Ear clinical symptoms | Day 0 and Day 6
  Evaluate ear-specific clinical symptoms (e.g. dryness and itchiness) through a MD questionnaire. This scale has been specifically developed for this clinical trial.
  - Clinical symptoms questionnaire (MD): Incidence of clinical symptoms and assessment scale of the intensity and frequency of the clinical symptoms (itchiness and dryness).
Patient clinical symptoms | Day 0 and Day 6
  Patient Questionnaire collecting clinical symptom prior and post-treatment This scale has been specifically developed for this clinical trial.
  - Clinical symptoms questionnaire (patient): Incidence of clinical symptoms and assessment scale of the intensity and frequency of the clinical symptoms (itchiness and dryness).
SAEs and AEs reported | Day 12
  Adverse Events (AEs) and Serious Adverse Events (SAEs) post-treatment.
Patient clinical symptom and ease-of-use | Day 6
  Patient Questionnaire assessing the ease-of-use of the medical device (Earol). This scale has been specifically developed for this clinical trial.
  - Ease of use of the device questionnaire: rating scale 0 - 10

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Clínica Universidad de Navarra, Madrid
  - Hospital QuironSalud Madrid, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital QuironSalud Marbella, Marbella
  - Hospital Quirónsalud Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Undecided